CLINICAL TRIAL: NCT00863187
Title: Assessing Antibody Responsiveness to Hepatitis B Vaccine in Aged Lymphoma Patients Undergoing Treatment With Rituximab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: doron melamed, technion
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 3097
Record Dates: First submitted 2009-02-15; First posted 2009-03-17 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-02

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab (Experimental): b cell depletion drug
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — b cell depletion

SUMMARY:
Background:

The ability of the immune system to function declines with aging. This is reflected by a marked decrease in the responsiveness to vaccinations and to infectious agents. Consequentially, there is a profound reduction in the quality of live and an increased dependency on the health systems. Studies have shown that the production of B lymphocytes in the bone marrow declines with aging and long-lived B cells accumulate in the periphery. Thus, instead of a juvenile repertoire of B cells that is capable to recognize any new pathogen, the repertoire of the elderly becomes more restricted and fails to respond to new antigens.

Working hypothesis and aims: We hypothesize that the dramatic change in the cellular composition in aging reflects homeostasis pressures that are set by long-lived peripheral B cells. Here, the investigators hypothesize that altering the homeostasis, by active depletion of the peripheral B cells, will revive B lymphopoiesis in the BM and rejuvenate the peripheral repertoire of B cells in aging. Consequentially, this will significantly improve immune responsiveness of aged individuals to new antigenic challenges.

Methods:

The investigators propose a parallel study in human and mouse. For our clinical study we will use old lymphoma patients that were treated with the B cell depleting therapy, RITUXIMAB, for transient B cell depletion and established full B cell reconstitution. We will test the responsiveness of these patients to hepatitis B vaccine and compare it to aged-matched control group. The investigators will also use old human CD20 transgenic mice where B cell depletion is imposed by anti human CD20 antibodies. In these experiments we will study physiological and immunological changes to understand aging mechanisms in the B lineage.

Expected results: We expect that old patients treated for B cell depletion will have an increased responsiveness to the hepatitis B vaccine relative to the control group.

Importance:

The investigators propose an efficient approach to improve immune response in the elderly population. This will increase efficacy of vaccination, reduce morbidity and improve quality of life. It will also reduce the cost of medical treatment. In addition, this study will show that senescence in the B lineage can be reversed, which is in contrast to the general concepts of aging.

Probable implications to the welfare and health of the aged population Medicine:

Improving the immune competence will increase efficacy of vaccination, reduce morbidity, and reduce dependency on health systems. This will significantly improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 55 years and older
* lymphoma
* rituximab

Exclusion Criteria:

* disease remission

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
anti hepatitis B antibodies | 3 month

SECONDARY OUTCOMES:
B cell proliferation and antibody secretion in response to stimulation in vitro | 3 month

REFERENCES:
- [Derived] Dowery R, Benhamou D, Benchetrit E, Harel O, Nevelsky A, Zisman-Rozen S, Braun-Moscovici Y, Balbir-Gurman A, Avivi I, Shechter A, Berdnik D, Wyss-Coray T, Melamed D. Peripheral B cells repress B-cell regeneration in aging through a TNF-alpha/IGFBP-1/IGF-1 immune-endocrine axis. Blood. 2021 Nov 11;138(19):1817-1829. doi: 10.1182/blood.2021012428. PMID 34297797